CLINICAL TRIAL: NCT01263301
Title: Differential Diagnosis for the Causes of Subclavian Steal for Patients With Vascular Access in the Forearm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mennonite Christian Hospital (Other)
Responsible Party: Principal Investigator, Ling-Chih, Wu, doctor, Mennonite Christian Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-06-024-ER
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2013-02-01 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Subclavian Steal
Keywords: subclavian steal; carotid duplex; subclavian stenosis; hemodialysis with vascular access in the upper limbs; the focus of this study is to see if duplex can be used as an tool to differentiate the different causes of subclavian steal syndromes
MeSH Terms: conditions — Subclavian Steal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- carotid duplex for hemolytic patients wtih SSS (Active Comparator): assigned intervention:carotid duplex
  Interventions: Device: carotid duplex
- carotid duplex for nonhemolytic patients with SSS (Active Comparator)
  Interventions: Device: carotid duplex

INTERVENTIONS:
Device: carotid duplex — Carotid duplex in the differential diagnosis of subclavian steal syndrome due to Arteriovenous Hemodialysis access in the Ipsilateral arm
  Other Names: steal syndrome

SUMMARY:
Subclavian steal phenomenon is normally observed in patients with stenosis of subclavian artery proximal to orifice of vertebral artery(V0). However, uremic patients undergoing hemodialysis using vascular access in the arm or forearm may also develop dialysis associated steal syndrome(DASS).For patients with symptomatic subclavian steal phenomenon, the treatment for these two groups is different. The investigators want to see if the investigators can use noninvasive duplex examination instead of invasive conventional angiography to do the differential diagnosis.

DETAILED DESCRIPTION:
Carotid duplex is widely used for diagnosis of subclavian steal syndrome. We have a patient who suffered from acute brain stem stroke after receiving hemodialysis for months. He has DM related uremia and the vascular access is in the forearm. Subclavian steal was found on duplex in the same arm for hemodialysis. We used standard cuff test for diagnosis of subclavian steal by carotid duplex examination. Accidentally, we found the flow of subclavian artery was back to normal when the cuff is on that stops the flow. We want to see if this phenomenon can be used to serve as a differential diagnostic tool for differentiation of subclavian steal caused by stenosis of subclavian artery or due to DASS.

ELIGIBILITY:
Inclusion Criteria:

* patients who revealed subclavian steal in the duplex study

Exclusion Criteria:

* patients who has vascular access in the arm instead of the forearm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: lingchih wu, Principal Investigator — Mennonite Christian Hospital
Locations (1):
- Mennonite Christial Hospital, Hualien City, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: enroll patients from Dec 2010 to July 2011. all enrolled patients have been studied by carotid duplex in Mennonite Christian hospital.
Pre-assignment Details: one patient with vascular access has been ruled out after enrollment for the subclavian artery revealed normal blood flow in duplex.
Groups:
- Carotid Duplex for Nonhemidialytic Patients Wtih SSS: using carotid duplex to study vertebral and subclavian artery, using cuff test to see the difference of flow during and after occlusion of blood vessel in the arm by cuff test for patients in the two groups
- Carotid Duplex for Hemodialytic Patients: After receiving written consent from patients with vascular access in the forearm, carotid duplex was done to especially see the flow pattern and direction of vertebral artery and subclavian artery in the ipsilateral side of vascular access.
  However, before carotid duplex, we didn't know which patients will show SSS.All 11 hemodialytic patients completed the study but only 2 showed the results of SSS. And for further analysis, we used these only 2.
Period: Overall Study
Arm/Group | Carotid Duplex for Nonhemidialytic Patients Wtih SSS | Carotid Duplex for Hemodialytic Patients
Started | 5 | 11
Completed | 5 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 11 hemodialytic patients particitated the study, only 2 shows SSS in carotid duplex. We analysed these 2 patients only.
Groups:
- Carotid Duplex for Nonhemodialytic Patients Wtih SSS: using carotid duplex (with cuff test) to study vertebral and subclavian artery to see the difference of flow during and after occlusion of blood vessel in the arm by cuff test
- Carotid Duplex for Hemodialytic Patients With SSS: After receiving written consent from patients with vascular access in the forearm, carotid duplex was done to especially see the flow pattern and direction of flow of vertebral artery and subclavian artery in the ipsilateral side of vascular access during and after the stop of flow in the arm by cuff test.
- Total: Total of all reporting groups
Arm/Group | Carotid Duplex for Nonhemodialytic Patients Wtih SSS | Carotid Duplex for Hemodialytic Patients With SSS | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.53) | 52.5 (0.70) | 59.71 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Taiwan | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change of Subclavian Flow to Normal Flow Pattern During Cuff Test
Description: we used carotid duplex duplex to study the change of subclavian arterial flow during cuff test to see if there is any difference between normal participants and patients under hemodialysis. There are two patterns seen. One is that the subclavian arterial flow reversed to normal flow pattern during cuff test. The other is that there is no change of subclavian flow pattern when the flow is stopped in the arm by cuff test.
Time Frame: two years
Population: for there are not too many patients who have subclavian steal found by carotid duplex, we just collected all patients during the study period that have subclavian steal and all patients with vascular access that signed written consent for the examination.
Measure: Number; unit: participants
Groups:
- Normal Parcipitants With Subclavian Steal: we use carotid duplex to study subclavian arterial flow before and during cuff test that stopped the flow in arm to see how many normal patients without vascular access will have subclavian arterial flow reversed to normal during the test
- Hemodialytic Patients With Subclavian Steal: we use carotid duplex to study subclavian arterial flow before and during cuff test that stopped the flow in arm to see how many patients with vascular access will have subclavian arterial flow reversed to normal pattern during the test
Arm/Group | Normal Parcipitants With Subclavian Steal | Hemodialytic Patients With Subclavian Steal
Number analyzed (Participants) | 5 | 2
participants | 0 | 2

2. Primary Outcome: no Change of Subclavian Arterial Flow During Cuff Test
Description: as for outcome 1
Time Frame: one year
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Normal Parcipitants With Subclavian Steal: we use carotid duplex to study subclavian arterial flow before and during cuff test that stopped the flow in arm to see how many normal patients without vascular access will have subclavian arterial flow remained unchanged during the cuff test
- Hemodialytic Patients With Subclavian Steal: we use carotid duplex to study subclavian arterial flow before and during cuff test that stopped the flow in arm to see how many patients with vascular access will have subclavian arterial flow remained unchanged during the cuff test
Arm/Group | Normal Parcipitants With Subclavian Steal | Hemodialytic Patients With Subclavian Steal
Number analyzed (Participants) | 5 | 2
participants | 5 | 0

3. Primary Outcome: Change of Vertebral Flow to Normal Flow Pattern During Cuff Test
Description: we used carotid duplex duplex to study the change of vertebral arterial flow during cuff test to see if there is any difference between normal participants and patients under hemodialysis. There are two patterns seen. One is that the vertebral arterial flow reversed to normal flow pattern during cuff test. The other is that there is no change of vertebral flow pattern when the flow is stopped in the arm by cuff test.
Time Frame: two year
Population: determined as above explained
Measure: Number; unit: participants
Groups:
- Normal Parcipitants With Subclavian Steal: we use carotid duplex to study vertebral arterial flow before and during cuff test that stopped the flow in arm to see how many normal patients without vascular access will have vertebral arterial flow reversed to normal during the test
- Hemodialytic Patients With Subclavian Steal: we use carotid duplex to study vertebral arterial flow before and during cuff test that stopped the flow in arm to see how many patients with vascular access will have vertebral arterial flow reversed to normal pattern during the test
Arm/Group | Normal Parcipitants With Subclavian Steal | Hemodialytic Patients With Subclavian Steal
Number analyzed (Participants) | 5 | 2
participants | 0 | 2

4. Primary Outcome: no Change of Vertebral Arterial Flow During Cuff Test
Description: as for outcome 3
Time Frame: 2 years
Population: as above explained
Measure: Number; unit: participants
Groups:
- Normal Parcipitants With Subclavian Steal: we use carotid duplex to study vertebral arterial flow before and during cuff test that stopped the flow in arm to see how many normal patients without vascular access will have vertebral arterial flow remained unchanged during the test
- Hemodialytic Patients With Subclavian Steal: we use carotid duplex to study vertebral arterial flow before and during cuff test that stopped the flow in arm to see how many patients with vascular access will have vertebral arterial flow remained unchanged during the test
Arm/Group | Normal Parcipitants With Subclavian Steal | Hemodialytic Patients With Subclavian Steal
Number analyzed (Participants) | 5 | 2
participants | 5 | 0

ADVERSE EVENTS:
Arm/Group | Carotid Duplex for Nonhemodialytic Patients Wtih SSS | Carotid Duplex for Hemodialytic Patients With SSS
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/11
Other Adverse Events (participants affected / at risk) | 0/5 | 0/11

LIMITATIONS AND CAVEATS:
the number of the study is small, no standard technique for measurement of blood flow of vascular access

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No